CLINICAL TRIAL: NCT05335304
Title: The Effects of Kinesio Taping, Rigid Taping, Thoracic Mobilization and Core Stabilization Approaches on Respiratory Muscle Morphology, Respiratory Muscle Strength, Exercise Capacity and Quality of Life in Stable COPD Patients.
Brief Title: The Effects of Different Physiotherapy Approaches in Stable COPD Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Emine Korkmaz, physiotherapist, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: physiotherapy approaches
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: COPD
Keywords: Taping, Muscle morphology, COPD, Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only the investigator who perform muscle thickness and muscle morphology measurements is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- intervention group 1 (Active Comparator): Kinesio taping and standard treatment program
  Interventions: Other: intervention group 1; Other: Pulmonary Rehabilitation
- intervention group 2 (Active Comparator): Rigid taping and standard treatment program
  Interventions: Other: intervention group 2; Other: Pulmonary Rehabilitation
- intervention group 3 (Active Comparator): Thoracic Mobilization and standard treatment program
  Interventions: Other: intervention group 3; Other: Pulmonary Rehabilitation
- intervention group 4 (Active Comparator): Core Stabilization and standard treatment program
  Interventions: Other: intervention group 4; Other: Pulmonary Rehabilitation
- Control group (Other): No intervention, only standard treatment program
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: intervention group 1 — Kinesio taping The intervention of this experimental study is therapeutic taping (kinesio tape) on the respiratory muscles of the participants.
  Arms: intervention group 1
Other: intervention group 2 — Rigid taping The intervention of this experimental study is therapeutic taping (rigid tape) on the respiratory muscles of the participants.
  Arms: intervention group 2
Other: intervention group 3 — Thoracic Mobilization The intervention of this experimental study is active-passive Thoracic mobilization techniques on the on the upper, middle or lower parts of the chest of the participants
  Arms: intervention group 3
Other: intervention group 4 — Core Stabilization The intervention of this experimental study is Core Stabilization exercises to the trunk muscles of the participants.
  Arms: intervention group 4
Other: Pulmonary Rehabilitation — Pulmonary Rehabilitation respiratory rehabilitation, stretching exercises, posture correction exercises

SUMMARY:
In our study, the effects of Kinesio Taping (KT), Rigid Taping (RT), Thoracic Mobilization (TM) and Core Stabilization (KS) approaches on respiratory muscle morphology, respiratory muscle strength, exercise capacity and quality of life will be examined in stable COPD patients. Study is designed as prospective, single-blinded, randomized-controlled study.

DETAILED DESCRIPTION:
The study is planned to compare the effects of different physiotherapy approaches on respiratory muscle morphology, respiratory muscle strength, exercise capacity and quality of life in stable COPD patients over 18 years of age.The study is carried out on 65 patients who applied to Muğla Training and Research Hospital with COPD patients. The patients are divided into 5 groups by randomization method. First group, Kinesio Taping group, inhibitory effect on upper trapezius and scalene muscles, facilitator effect on diaphragm and intercostal muscles will be applied. The second group, Rigid Taping group, inhibitory effect on upper trapezius and scalene muscles, facilitator effect on diaphragm and intercostal muscles will be applied. The third group,Thoracic Mobilization group, Modified Active-Passive Thoracic mobilization will be performed according to the patients' conditions. Thoracic Mobilization techniques will be used to improve thoracic mobility in the upper, middle or lower parts of the chest. The fourth group,In Core Stabilization group, five different trunk stabilization exercises will be performed. Fifth group is the control group and no taping was done. A standard treatment program is applied for the individuals in the whole group. Evaluations is made before and after treatment (3 and 6 weeks). Evaluation parameters is respiratory muscle morphology, respiratory muscle strength, exercise capacity and quality of life.

The respiratory muscle morphology is measured by the radiologist, and all other measurements and treatments were performed by the physiotherapist. Pulmonary function test will be measured using spirometry, respiratory muscle strength using mouth pressure device, functional exercise capacity using 6-minute walk test, quality of life using Leicester Cough Questionnaire, dyspnea using Modified Medical Research Council Dyspnea Scale and, symptoms using COPD Assessment Tests.

The data obtain from the research will be analyzed using the SPSS program. Statistical significance level will be accepted as p<0.05. In the statistical difference analysis between groups, one-way ANOVA test will be used for parametric data and Kruskal- Wallis test will be used for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

1. People with stable COPD,
2. Patients with spirometric measurements of GOLD 2-3 according to the new GOLD classification and A, B according to symptoms and exacerbations
3. To be 18 years or older,
4. No acute exacerbation in the last 3 weeks,
5. Alterations in medical treatment and not using any antibiotics in last 3 weeks,
6. Not being included in the pulmonary rehabilitation program in the last 6 months,
7. Volunteering to participate in study

Exclusion Criteria:

1. Orthopedic and neuromuscular disorders,
2. Advanced heart failure,
3. Aortic stenosis, deep vein thrombosis, pacemaker,
4. Patients with acute exacerbation of symptoms in the previous three weeks,
5. Those with weak cognitive function will be excluded from the study.
6. Patients who are unable to cooperate will also be considered ineligible.
7. Irritation, infection, allergic reaction, scarred burn or open wound around application area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle morphology | Change in muscle thickness at 6 week
  Respiratory muscle morphology measurement will be made by the radiologist with the US imaging method. It will be applied to the diaphragm, intercostal muscles, upper trapezius and scalene muscles.
Respiratory muscle strength | Change in MİP and MEP at 6 week
  Maximum inspiratory pressure (Pimax) and maximum expiratory pressure (PEmax) will be evaluated using an electronic pressure transducer.Measurements will be made according to the guidelines of the American Thoracic Society/European Respiratory Society.
  Pimax at residual volume and PEmax from Total lung capacity, Maximal inspiratory pressure will be determined by placing a nose clip instructed to exhale to residual volume followed by maximum inspiration.
  To assess maximal expiratory pressure, the patient is instructed to inhale until total lung capacity is reached, followed by a forced exhalation. Three evaluations will be recorded and the best value will be used.
6-minute walk test | Change in distance at 6 week
  It will be held in a 30 m barrier-free corridor. The measurement will be made according to the guidelines of the American Thoracic Society. The 6MWT will be repeated 2 times and the result will be given as a percentage of the predicted values. Patients will rest for 30 minutes between tests and the maximum distance will be recorded.
Leicester Cough Questionnaire | Change in quality of life at 6 week
  It consists of 19 items in 3 subcategories (physical, psychological, social) assessing the quality of life associated with chronic cough. Each question is evaluated using a 7-point Likert-type scoring system. The total score is obtained by summing the 3 sub-category scores. High scores are indicative of good quality of life.

SECONDARY OUTCOMES:
Modified Borg Scale | Change in dyspnea at 6 week
  It is a scale used to evaluate the severity of dyspnea on exertion and the severity of dyspnea at rest. It consists of ten items describing the severity of dyspnea according to their degrees. 0 scales as no dyspnea, 10 as very severe dyspnea
COPD Assessment Test (CAT) | Change in healty status at 6 week
  It was developed to measure the health status and to evaluate the disease effect and severity in COPD. The CAT consists of eight questions, covering problems such as shortness of breath, cough, sputum production, as well as symptoms such as fatigue and sleep problems. Perfect health: 0 points (minimum), worst health: 40 points. (max score)
Static and dynamic lung volumes Pulmonary Function Tests | Change in lung volumes at 6 week.
  In order to evaluate pulmonary functions, FVC, FEV1, FEV1/FVC, Peak flow rate (PEF), 25-75% (FEF 25-75%) flow rate of forced expiratory volume will be taken in sitting position according to ATS/ERS criteria. Pulmonary function test parameters will be expressed as a percentage of actual values and expected values.
Modified Medical Research Council | Change in perception of dyspnea at 6 week
  The dyspnea scale will be used to evaluate the severity of dyspnea during activities of daily living. It will be graded from 0 (absence of dyspnea during strenuous exercise) to 4 (dyspnea during daily activities). The dyspnea perception scale will be questioned to what extent the patients have perceived dyspnea in daily activities in the last week.
COPD and Asthma Fatigue Scale | Change in fatigue score at 6 week
  The original scale consists of 12 items and a Likert-type scale (1=never, 2=rarely, 3=sometimes, 4=often, 5=very often) is used for responses. Scoring of the scale is in a five-point Likert type and a total value between 12 and 60 points is obtained.
Posture analysis | Change in posture at 6 week
  "Posture Screen Mobile" mobile application will be used via smart phone to evaluate static posture.
Chest anterior-posterior diameter measurement | Change in chest diameter at 6 week
  Rib cage measurements Anterior and posterior diameter will be measured using a caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Baki Umut Tuğay, Study Chair — Muğla Sıtkı Koçman University

IPD SHARING:
Plan to Share IPD: No